CLINICAL TRIAL: NCT07180641
Title: REGISTRO NACIONAL DE METÁSTASIS HEPÁTICAS DE CÁNCER NO COLORRECTAL
Brief Title: National Registry of Hepatic Metastases From Non-Colorectal Cancer"
Acronym: REMENOCOR
Status: Completed | Type: Observational
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Other Study IDs: 2023.238
Record Dates: First submitted 2025-08-25; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Non-colorectal Liver Metastasis; Liver Metastasis; Non-neuroendocrine Liver Metastasis; Liver Metastases; Non-colorectal Liver Metastases; Non-neuroendocrine Liver Metastases; Liver Resection; Hepatectomy
Keywords: Non-colorectal non-neuroendocrine liver metastases; Liver metastases; Liver resection; Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with non-colorectal liver metastases: Patients who underwent liver resection for non-colorectal liver metastases from January 2010 to December 2022

SUMMARY:
The investigators designed this observational, retrospective, multicenter study including all patients who underwent surgery for non-colorectal liver metastases between January 2010 and December 2022, with the aim of establishing a series of recommendations for the treatment of liver metastases from various extrahepatic primary tumors

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for liver surgery due to non-colorectal liver metastases, regardless of the primary tumor origin, via open or minimally invasive approach

Exclusion Criteria:

* Patients undergoing surgery for colorectal liver metastases, emergency surgical interventions and patients younger than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for liver surgery due to non-colorectal liver metastases, regardless of the primary tumor origin, via open or minimally invasive approach, from January 2010 to December 2022
Sampling Method: Probability Sample
Enrollment: 1039 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 5 years from liver resection
  Time from the date of liver resection for non-colorectal metastases to death from any cause. Survival will be assessed for up to 5 years postoperatively
Progression-Free Survival | 5 years from surgery
  Time from the date of liver resection for non-colorectal metastases to the date of documented disease progression or death from any cause, whichever occurs first. Patients without progression or death will be censored at the last follow-up

SECONDARY OUTCOMES:
Postoperative Morbidity Rate | 90 days from surgery
  Incidence of any postoperative complications occurring within 90 days after liver resection, including but not limited to infections, bleeding, bile leaks, and other surgical complications, classified according to standard criteria.
Postoperative Mortality Rate | 90 days from surgery
  Proportion of patients who die from any cause within 90 days following liver resection surgery.
Recurrence Pattern | Up to 5 years from liver resection
  Distribution and characterization of tumor recurrence (hepatic, extrahepatic, or both) after liver resection for non-colorectal metastases.
Length of hospital stay | Perioperative/Periprocedural
  Number of days from surgery to discharge following liver resection
R0 Resection Rate | At surgery
  Proportion of patients achieving complete microscopic liver tumor resection (R0) during liver resection

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared with all investigators who have participated in this multicenter study and who have expressed interest in its follow-up and execution. The data will be shared anonymously, as each patient is assigned a unique anonymized identification number unrelated to their clinical records. Access to the data will be available for a period of five years following the end of recruitment, which was June 2025. There is no official repository; interested investigators must contact me directly, and I will provide them with unique and private access to the data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 5 years following the end of recruitment, which was June 2025
Access Criteria: All investigators who have participated in this multicenter study and who have expressed interest in its follow-up and execution.